CLINICAL TRIAL: NCT01123018
Title: Screening for Memory Studies
Status: Active, not recruiting | Type: Observational
Sponsor: John Wesson Ashford Jr (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, John Wesson Ashford Jr, Director, VA Palo Alto Health Care System
Organization: VA Palo Alto Health Care System (U.S. Federal Agency)
Other Study IDs: SU-06302009-2900
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Memory Loss; Memory Deficits; Dementia
Keywords: Memory Loss
MeSH Terms: conditions — Memory Disorders; Dementia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Older Adults: Persons over age 60 Participants will complete the Memtrax memory screening test
  Interventions: Behavioral: Memtrax Memory screening test

INTERVENTIONS:
Behavioral: Memtrax Memory screening test — Memory Screening test
  Other Names: Memory screening

SUMMARY:
We hope to recruit participants into various clinical trials and research projects.

DETAILED DESCRIPTION:
The purpose of this protocol is to advertise, recruit, and do a preliminary screen for various clinical trials. Anonymous information collected will be entered in a database available to researchers connected with the Stanford/VA Aging Clinical Research Center, located at VA Palo Alto Health Care System, Palo Alto Division.

ELIGIBILITY:
Inclusion Criteria:

* Age 55 or over.

Exclusion Criteria:

* Major psychiatric problems.
* Major medical problems.
* Aversion to test-taking.

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy older adults with memory concerns
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2007-06; Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: J. Wesson Ashford Jr., MD, PhD, Principal Investigator — Stanford University
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ashford JW, Borson S. Primary care screening for dementia and mild cognitive impairment. JAMA. 2008 Mar 12;299(10):1132-3; author reply 1133-4. doi: 10.1001/jama.299.10.1132-b. No abstract available. PMID 18334685